CLINICAL TRIAL: NCT01232569
Title: A Randomized, Double-blind, Parallel Group Study of Safety and the Effect on Clinical Outcome of Tocilizumab Subcutaneous (sc) Versus Placebo sc in Combination With Traditional Disease Modifying Anti-rheumatic Drugs (DMARDs) in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) Given Subcutaneously in Combination With Traditional DMARDs in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA25220; 2010-019912-18 (EudraCT Number)
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Tocilizumab 162 mg sc (Experimental): Patients will receive tocilizumab 162 mg subcutaneously (sc) every 2 weeks for 24 weeks.
  Interventions: Drug: Tocilizumab 162 mg
- Placebo sc (Placebo Comparator): Patients will receive placebo subcutaneously (sc) every 2 weeks for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab 162 mg — Tocilizumab will be supplied in a ready-to-use, single-use, pre-filled syringe. Patients and/or caregivers will be trained to administer the injection.
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab 162 mg sc
Drug: Placebo — Placebo will be supplied in a ready-to-use, single-use, pre-filled syringe. Patients and/or caregivers will be trained to administer the injection.
  Arms: Placebo sc

SUMMARY:
This randomized, parallel-group, placebo-controlled, multicenter study will evaluate the reduction in disease activity and the safety of tocilizumab (RoActemra/Actemra) in combination with traditional disease-modifying anti-rheumatic drugs (DMARDs) in patients with active, moderate to severe rheumatoid arthritis. In the double-blind part of the study, patients will be randomized to receive either 162 mg tocilizumab or placebo subcutaneously every 2 weeks for 24 weeks using a pre-filled syringe. In the open-label part of the study, patients will be randomized to receive 162 mg tocilizumab subcutaneously every 2 weeks from Week 24 to Week 96 using a pre-filled syringe or an auto-injector.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ years of age.
* Moderate to severe rheumatoid arthritis of ≥ 6 months duration.
* Receiving treatment on an outpatient basis.
* Swollen joint count (SJC) ≥ 6 (66 joint count) and tender joint count (TJC)≥ 8 (68 joint count) at screening and study start.
* On a stable dose of disease-modifying anti-rheumatic drugs for at least 8 weeks prior to study start.

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Rheumatic autoimmune disease other than rheumatoid arthritis, Secondary Sjögren's Syndrome with rheumatoid arthritis is allowed.
* Functional class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in Rheumatoid Arthritis.
* Diagnosis of juvenile idiopathic arthritis or juvenile rheumatoid arthritis and/or rheumatoid arthritis before the age of 16 years.
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis.
* History of malignancy, active or recurrent infections, positive to hepatitis B surface antigen or hepatitis C antibody, active tuberculosis, serious allergy to biologics, or a history of diverticular disease or other symptomatic GI conditions that might predispose to perforations.

Other inclusion and exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (118):
- United States (39):
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Fullerton, California
  - San Diego, California
  - San Leandro, California
  - West Hills, California
  - Trumbull, Connecticut
  - Boca Raton, Florida
  - Jupiter, Florida
  - Ormond Beach, Florida
  - Sarasota, Florida
  - Gainesville, Georgia
  - Idaho Falls, Idaho
  - Meridan, Idaho
  - Springfield, Illinois
  - Vernon Hills, Illinois
  - Crofton, Maryland
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Flowood, Mississippi
  - Jackson, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Brooklyn, New York
  - Belmont, North Carolina
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Wexford, Pennsylvania
  - Wyomissing, Pennsylvania
  - Memphis, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tacoma, Washington
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - San Miguel de Tucumán
- Australia (2):
  - Cairns
  - Kogarah
- Brazil (8):
  - Curitiba
  - Goiânia
  - Juiz de Fora
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - São Paulo
  - Vitória
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Canada (5):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - London, Ontario
  - Ottawa, Ontario
  - Pointe-Claire, Quebec
- Colombia (3):
  - Bogotá
  - Chia-cundinamarca
  - Medellín
- Greece (2):
  - Athens
  - Thessaloniki
- Guatemala City, Guatemala
- Hungary (2):
  - Budapest
  - Debrecen
- Israel (6):
  - Ashkelon
  - Beersheba
  - Haifa
  - Ramat Gan
  - Rishon LeZiyyon
  - Tel Aviv
- Malaysia (3):
  - Batu Caves
  - Kota Kinabalu
  - Kuala Lumpur
- Mexico (10):
  - Chihuahua City
  - Culiacán
  - Guadalajara
  - León
  - Mexicali
  - Mérida
  - México
  - Morelia
  - Obregón
  - Querétaro
- Otahuhu, New Zealand
- Panama City, Panama
- Philippines (3):
  - Cebu
  - Davao City
  - Manila
- Poland (7):
  - Bytom
  - Działdowo
  - Elblag
  - Kościan
  - Krakow
  - Torun
  - Warsaw
- Russia (8):
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Ufa
  - Voronezh
- South Africa (3):
  - Durban
  - Pinelands
  - Pretoria
- Spain (3):
  - A Coruña
  - Oviedo
  - Seville
- Switzerland (4):
  - Fribourg
  - Geneva
  - Lausanne
  - Zurich
- Bangkok, Thailand

REFERENCES:
- [Derived] Kivitz A, Olech E, Borofsky M, Zazueta BM, Navarro-Sarabia F, Radominski SC, Merrill JT, Rowell L, Nasmyth-Miller C, Bao M, Wright S, Pope JE. Subcutaneous tocilizumab versus placebo in combination with disease-modifying antirheumatic drugs in patients with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2014 Nov;66(11):1653-61. doi: 10.1002/acr.22384. PMID 24942540

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 656 patients randomized into the study (437 to the tocilizumab arm and 219 to the placebo arm), 438 patients received tocilizumab as their first dose and 218 received placebo as their first dose because of a dose administration error with 1 patient.
Groups:
- Tocilizumab 162 mg sc - Double-blind Treatment Period: Patients received tocilizumab 162 mg subcutaneously (sc) every 2 weeks for 24 weeks.
- Placebo sc - Double-blind Treatment Period: Patients received placebo sc every 2 weeks for 24 weeks.
- Tocilizumab Pre-filled Syringe - Open-label Extension Period: Patients received tocilizumab 162 mg sc via a pre-filled syringe every 2 weeks for 72 weeks.
- Tocilizumab Auto-injector - Open-label Extension Period: Patients received tocilizumab 162 mg sc via auto-injector every 2 weeks for 72 weeks.
Period: Double-blind Treatment Period
Arm/Group | Tocilizumab 162 mg sc - Double-blind Treatment Period | Placebo sc - Double-blind Treatment Period | Tocilizumab Pre-filled Syringe - Open-label Extension Period | Tocilizumab Auto-injector - Open-label Extension Period
Started | 438 | 218 | 0 (There were no participants in this reporting group in this period.) | 0 (There were no participants in this reporting group in this period.)
Completed | 410 | 209 | 0 | 0
Not Completed | 28 | 9 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 0 | 0
Not completed — Escape | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Adverse Event (Except Anaphylaxis) | 9 | 3 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Period: Open-label Extension Period
Arm/Group | Tocilizumab 162 mg sc - Double-blind Treatment Period | Placebo sc - Double-blind Treatment Period | Tocilizumab Pre-filled Syringe - Open-label Extension Period | Tocilizumab Auto-injector - Open-label Extension Period
Started | 0 (There were no participants in this reporting group in this period.) | 0 (There were no participants in this reporting group in this period.) | 230 (Some participants who completed the double-blind period did not enter the open-label period.) | 227 (Some participants who completed the double-blind period did not enter the open-label period.)
Completed | 0 | 0 | 203 | 200
Not Completed | 0 | 0 | 27 | 27

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics are reported for the safety population which included all patients who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. One patient who received tocilizumab had no post-baseline safety data and was excluded from the safety population.
Groups:
- Tocilizumab 162 mg sc: Patients received tocilizumab 162 mg subcutaneously (sc) every 2 weeks for 24 weeks.
- Placebo sc: Patients received placebo subcutaneously (sc) every 2 weeks for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 162 mg sc | Placebo sc | Total
Number analyzed (Participants) | 437 | 218 | 655
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.49) | 52.0 (11.67) | 52.1 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 180 | 555
  Male | 62 | 38 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an American College of Rheumatology 20 (ACR20) Response at Week 24
Description: A patient had an ACR20 response if there was at least a 20% improvement, ie, reduction from baseline, in tender and swollen joint counts (28 assessed joints) and in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, left end=no disease activity [symptom-free and no arthritis symptoms], right end=maximum disease activity; patient assessment of pain in previous 24 hours on a VAS (left end=no pain and right end=unbearable pain); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and acute-phase reactant (either C-reactive protein or erythrocyte sedimentation rate).
Time Frame: Baseline to Week 24
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug. Patients were assigned to the ITT population as randomized, irrespective of the treatment actually received. Only patients with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 437 | 219
Percentage of patients | 60.9 [56.3 to 65.4] | 31.5 [25.4 to 37.7]
Statistical Analysis 1: Comparison: Tocilizumab 162 mg sc vs Placebo sc; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Analysis adjusted for the randomization stratification factors applied at Baseline (region and weight category); Mean Difference (Final Values) = 29.5, 95% CI 2-sided [22.0 to 37.0]

2. Secondary Outcome: Percentage of Patients With ACR50 and ACR70 Responses at Week 24
Description: A patient had an ACR50 response if there was at least a 50% improvement in the ACR scores. A patient had an ACR70 response if there was at least a 70% improvement in the ACR scores.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 437 | 219
Percentage of patients
  ACR50 | 39.8 [35.2 to 44.4] | 12.3 [8.0 to 16.7]
  ACR70 | 19.7 [16.0 to 23.4] | 5.0 [2.1 to 7.9]

3. Secondary Outcome: Time to Onset of ACR20, ACR50, and ACR70 Responses
Description: Time to first ACR response was calculated as the number of days between the date of the first ACR response minus the date of the first dose of study drug. Median days are reported.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 437 | 219
Days
  ACR20 | 57 [57 to 58] | 86 [85 to 113]
  ACR50 | 115 [113 to 141] | NA [NA to NA] — Not calculable due to too few events.
  ACR70 | 174 [172 to NA] — Not calculable due to too few events. | NA [NA to NA] — Not calculable due to too few events.

4. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Week 24
Description: Joints (28 joints) will be assessed and classified as swollen/not swollen and tender/not tender by pressure and joint manipulation on physical examination.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 432 | 219
Joint count
  Tender Joint Count | -14.8 (15.0) | -8.1 (14.2)
  Swollen Joint Count | -9.6 (9.7) | -5.9 (10.2)

5. Secondary Outcome: Change From Baseline in C-reactive Protein at Week 24
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 345 | 124
mg/dL | -1.7 (2.6) | -0.1 (1.8)

6. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate at Week 24
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 347 | 124
mm/hr | -36.4 (23.6) | -9.5 (22.7)

7. Secondary Outcome: Change From Baseline in the Patient's and the Physician's Global Assessment of Disease Activity Visual Analog (VAS) Score
Description: Patients and physicians assessed the patient's disease activity in the previous 24 hours on a 100 mm visual analog scale, where the extreme left end of the line represented "no disease activity" (symptom-free and no arthritis symptoms) and the extreme right end represented "maximum disease activity". Scores ranged from 0 to 100 with a higher score indicating more disease activity. A negative change score indicated less disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 348 | 124
Units on a scale
  Patient's Global Assessment VAS, N=346, 123 | -32.0 (27.6) | -20.9 (25.2)
  Physician's Global Assessment VAS, N=348, 124 | -36.9 (22.5) | -30.7 (25.8)

8. Secondary Outcome: Change From Baseline in the Patient's Pain Visual Analog Score
Description: Patients assessed their pain in the previous 24 hours on a visual analog scale, where the extreme left end of the line represented "no pain" and the extreme right end represented "unbearable pain". Scores ranged from 0 to 100 with a higher score indicating more pain. A negative change score indicated less pain.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 346 | 123
Units on a scale | -28.1 (27.2) | -15.0 (28.3)

9. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: The HAQ-DI is a questionnaire specific for rheumatoid arthritis and consists of 20 questions referring to 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Patients completed the questionnaire by answering the 20 questions on a scale of 0 (without difficulty) to 3 (unable to do). The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 348 | 124
Units on a scale | -0.5 (0.6) | -0.3 (0.6)

10. Secondary Outcome: Percentage of Patients With an Improvement of ≥ 0.3 Units From Baseline in the HAQ-DI Score at Week 24
Description: as for outcome 9
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 348 | 124
Percentage of patients | 58.0 [52.9 to 63.2] | 46.8 [38.0 to 55.6]

11. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) at Week 24
Description: The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 344 | 123
Units on a scale | -3.3 (1.4) | -1.8 (1.3)

12. Secondary Outcome: Percentage of Patients With a DAS28 Score ≤ 3.2 (DAS28 Low Disease Activity) at Week 24
Description: as for outcome 11
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 347 | 124
Percentage of patients | 45.2 [40.0 to 50.5] | 15.3 [9.0 to 21.7]

13. Secondary Outcome: Percentage of Patients With a DAS28 Score < 2.6 (DAS28 Remission) at Week 24
Description: as for outcome 11
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 347 | 124
Percentage of patients | 32.0 [27.1 to 36.9] | 4.0 [0.6 to 7.5]

14. Secondary Outcome: Percentage of Patients With Good, Moderate, or no European League Against Rheumatism (EULAR) Responses at Week 24
Description: Change of the Disease Activity Score 28 score from baseline was used to determine EULAR responses of good, moderate, or no response. For a post-baseline score ≤ 3.2, a change from baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-baseline score > 3.2 to ≤ 5.1, a change from baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-baseline score > 5.1, a change from baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-baseline scores > 3.2.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 374 | 138
Percentage of patients
  Good Response | 41.7 | 13.8
  Moderate Response | 44.9 | 54.3
  No Response | 13.4 | 31.9

15. Secondary Outcome: Change From Baseline in the Van Der Heijde Modified Sharp Radiographic Score at Week 24
Description: The degree of joint damage was assessed using the van der Heijde modified total Sharp score (mTSS). The methodology quantifies the extent of bone erosions for 44 joints and joint space narrowing (JSN) for 42 joints, with higher scores representing greater damage. The independent read of X-ray images was performed by 2 primary readers. In case of discrepancy between the 2 primary readers, an adjudicator was involved. The mTSS can range from 0 to 448 with a higher score indicating more joint damage. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 391 | 186
Units on a scale | 0.62 (2.692) | 1.23 (2.816)

16. Secondary Outcome: Change From Baseline in the Physical and Mental Component Scores of the Short Form 36 (SF-36) Health Survey at Week 24
Description: The SF-36 Health Survey uses patient-reported symptoms on 8 subscales to assess health-related quality of life (HRQoL). The Physical Component Summary (PCS) score summarizes the subscales Physical Functioning, Role-Physical, Bodily Pain, and General Health. The Mental Component Summary (MCS) score summarizes the subscales Vitality, Social Functioning, Role-Emotional, and Mental Health. Each score was scaled from 0 to 100 with a higher score indicating better HRQoL. A positive change score indicates an improvement in HRQoL.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 347 | 123
Units on a scale
  Physical Component | 7.2 (8.0) | 4.3 (5.9)
  Mental Component | 6.1 (10.8) | 3.0 (9.7)

17. Secondary Outcome: Change From Baseline in Hemoglobin at Week 24
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tocilizumab 162 mg sc | Placebo sc
Number analyzed (Participants) | 343 | 123
g/L | 11.0 (12.6) | 0.0 (7.1)

ADVERSE EVENTS:
Description: Safety population: All patients who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. One patient who received tocilizumab had no post-baseline safety data and was excluded from the safety population.
  Due to the study design, some participants received tocilizumab throughout the study, others not.
Groups:
- Tocilizumab Pre-filled Syringe: Patients received tocilizumab 162 mg sc via a pre-filled syringe every 2 weeks for 24 weeks. In addition, this reporting group includes participants re-randomized at Week 24 to tocilizumab 162 mg sc via a pre-filled syringe every 2 weeks for 72 weeks (Weeks 25-96).
- Placebo Pre-filled Syringe: Patients received placebo subcutaneously (sc) via a pre-filled syringe every 2 weeks for 24 weeks.
- Tocilizumab Pre-filled Syringe to Tocilizumab Auto-injector: Patients received tocilizumab 162 mg sc via a pre-filled syringe every 2 weeks for 24 weeks followed by tocilizumab162 mg sc via an autoinjector every 2 weeks for 72 weeks.
- Placebo Pre-filled Syringe to Tocilizumab Pre-filled Syringe: Patients received placebo sc via a pre-filled syringe every 2 weeks for 24 weeks followed by tocilizumab162 mg sc via a pre-filled syringe every 2 weeks for 72 weeks.
- Placebo Pre-filled Syringe to Tocilizumab Autoinjector: Patients received placebo sc via a pre-filled syringe every 2 weeks for 24 weeks followed by tocilizumab162 mg sc via an autoinjector every 2 weeks for 72 weeks.
Arm/Group | Tocilizumab Pre-filled Syringe | Placebo Pre-filled Syringe | Tocilizumab Pre-filled Syringe to Tocilizumab Auto-injector | Placebo Pre-filled Syringe to Tocilizumab Pre-filled Syringe | Placebo Pre-filled Syringe to Tocilizumab Autoinjector
Serious Adverse Events (participants affected / at risk) | 36/437 | 8/218 | 17/168 | 2/61 | 0/59
Other Adverse Events (participants affected / at risk) | 212/437 | 65/218 | 89/168 | 35/61 | 33/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Pre-filled Syringe (N=437) | Placebo Pre-filled Syringe (N=218) | Tocilizumab Pre-filled Syringe to Tocilizumab Auto-injector (N=168) | Placebo Pre-filled Syringe to Tocilizumab Pre-filled Syringe (N=61) | Placebo Pre-filled Syringe to Tocilizumab Autoinjector (N=59)
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Joint abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ludwig angina (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhagic inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Adrenocortical insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Pre-filled Syringe (N=437) | Placebo Pre-filled Syringe (N=218) | Tocilizumab Pre-filled Syringe to Tocilizumab Auto-injector (N=168) | Placebo Pre-filled Syringe to Tocilizumab Pre-filled Syringe (N=61) | Placebo Pre-filled Syringe to Tocilizumab Autoinjector (N=59)
Alanine aminotransferase increased (Investigations) | 67 | 13 | 24 | 6 | 10
Aspartate aminotransferase increased (Investigations) | 40 | 10 | 14 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 52 | 14 | 21 | 12 | 6
Headache (Nervous system disorders) | 28 | 13 | 8 | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 25 | 1 | 8 | 5 | 7
Nasopharyngitis (Infections and infestations) | 35 | 5 | 16 | 5 | 4
Urinary tract infection (Infections and infestations) | 26 | 7 | 15 | 2 | 4
Sinusitis (Infections and infestations) | 13 | 1 | 8 | 5 | 1
Bronchitis (Infections and infestations) | 13 | 2 | 4 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 21 | 3 | 6 | 3 | 5
Gastritis (Gastrointestinal disorders) | 6 | 3 | 1 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 13 | 1 | 5 | 0 | 3
Hypertension (Vascular disorders) | 26 | 8 | 9 | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 | 2 | 5 | 2 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 2 | 2 | 6 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 14 | 4 | 12 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.